CLINICAL TRIAL: NCT05647434
Title: Effect of Sustained Inflations on Lung Atelectasis During Pediatric Laparoscopic Surgery as Determined by Lung Ultrasound: a Randomized Controlled Trial
Brief Title: Effect of Sustained Inflations on Lung Atelectasis During Pediatric Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hussein Sayed Hasan, lecturer of anesthesia , surgical ICU and pin managment, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD-240-2021
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Ventilator Lung

STUDY DESIGN:
Who Masked: Investigator
Masking Description: lung ultrasound will be done by same doctor in both groups who is trained in lung ultrasound he will enter operating room only during ultrasound examination. not to know sustained inflations done in which cases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group C (No Intervention): conventional ventilation
- group SI (Active Comparator): Sustained inflations done after ultrasound during capnoperitoneum every 20 min.
  Interventions: Procedure: sustained inflations

INTERVENTIONS:
Procedure: sustained inflations — Sustained inflation will be applied at a pressure of 30 cmH2O and will be held for a period of 30 secs. After each SI the standard ventilatory settings will be resumed with a PEEP setting of 8 cmH2O to prevent lung derecruitment. Lung recruitment will be stopped immediately if mean arterial pressure and/or heart rate change by at least 25% from baseline values.
  Arms: group SI

SUMMARY:
The aim of our study is to assess the beneficial effect of sustained inflations as a recruitment manoeuvre, using LUS examinations, on the degree of lung atelectasis that occurs in pediatric patients undergoing laparoscopic surgery.

Objectives

* To assess the effect of general anaesthesia and capnoperitoneum on lung atelectasis in the paediatric patients by using LUS examination
* To assess the effect of sustained inflations as a recruitment manoeuvre in decreasing lung atelectasis caused by general anaesthesia and capnoperitoneum by using LUS examination

Hypothesis Our main hypothesis is that the use of repeated Sustained Inflation as a recruitment manoeuvre in pediatric patients undergoing laparoscopic surgery will result in decreased atelectasis compared to conventional ventilation.

DETAILED DESCRIPTION:
Our study will be conducted in Cairo University Specialized Pediatric Hospital (Abo El Reesh Hospital), after approval of the research ethical committee. An informed signed parental consent will be obtained from all study participants before their enrolment in the study. recruitment of cases will be started after registration in clinicaltrials.gov and getting unique number

Methodology

* Study Design Prospective Randomised Controlled Study

  * Study Setting and Location The study will be conducted in the operating theatres at Cairo University Specialized Pediatric Hospital (Abo El Rich Hospital), Faculty of Medicine, Cairo University.

    * Study Population 40 pediatric patients undergoing laparoscopic surgery will be included in the study. The patients will be randomly allocated into one of the two study groups; 20 patients per group.

      1. Study protocol Following approval from anesthesia department's ethics and research committee, all patients fulfilling the eligibility criteria will be enrolled in the study. An informed signed parental consent will be obtained.

         Anesthesia Standard ECG, noninvasive blood pressure measurement, time-based capnography and pulse oximetry will be used as monitors. Anesthesia will be induced with Sevofluorane using a Mapelson E (modification of Ayre's T-piece) circuit. An Intravenous access will be obtained. Fentanyl 2 μg/kg and Atracurium 0.5 mg/kg will be administered intravenously before intubation with a cuffed endotracheal tube of appropriate size followed by controlled ventilation. The lungs will be ventilated in a volume control mode using a FiO2 of 0.5, a tidal volume of 6 ml/kg, a positive end-expiratory pressure (PEEP) of 5 cmH2O, an inspiratory: expiratory ratio of 1:2, respiratory rate between 20 and 30 breaths per minute to maintain end tidal CO2 between 30-35 mmHg. Anesthesia will be maintained with sevoflurane 2% in the supine position. Top up doses of muscle relaxant will be administered as needed.

         Randomisation The patients will be randomly allocated. The randomization sequence will be concealed in sealed opaque envelopes.

         • Control group (C-group): patients will receive the conventional ventilatory settings as described above.
         * Sustained inflation group (SI group): After induction of capnoperitoneum, LUS examination will be performed. Sustained inflation will be performed immediately after this LUS examination, and will be repeated every 20 minutes during the period of capnoperitoneum. Sustained inflation will be applied at a pressure of 30 cmH2O and will be held for a period of 30 secs. After each SI the standard ventilatory settings will be resumed with a PEEP setting of 8 cmH2O to prevent lung derecruitment. Lung recruitment will be stopped immediately if mean arterial pressure and/or heart rate change by at least 25% from baseline values.

         Lung Ultrasound LUS will be performed using the SonoSite M Turbo (USA) with a linear multi-frequency 6-13 MHz probe. Each hemithorax will be divided into six regions, using three longitudinal lines (parasternal, anterior and posterior axillary) and two axial lines (one above the diaphragm and the other 1 cm above the nipples). The 12 lung regions will be scanned sequentially from right to left, cranial to caudal and anterior to posterior. Each region will be assessed using a two dimensional view with the probe placed parallel to the ribs. In general, the posterior areas are those with the highest incidence of anesthesia-induced atelectasis. (30) An aeration score previously described for adults will be applied in our pediatric patients. (27) Four LUS patterns were defined according to the degree of B lines: (0) fewer than three isolated B lines; (1) multiple well defined B lines; (2) multiple coalescent B lines and (3) white lung. The sum of the points obtained in all the 12 lung areas will constitute the lung aeration score, ranging from 0-36 for the whole thorax. This score is inversely proportional to the degree of lung aeration and directly proportional to the degree of lung atelectasis. (30)

         Patients will be studied at three points:
         * Before capnoperitoneum: 5 minutes after induction of anaesthesia, baseline recordings will be obtained.
         * During capnoperitoneum: measurements will be performed 10 minutes after starting the capnoperitoneum.
         * After capnoperitoneum: 5 minutes after the end of surgery.
      2. Measurement tools

         • Lung aeration score.

         • Hemodynamic parameters: HR, Non-invasive blood pressure, end-tidal CO2 and oxygen saturation.

         • Respiratory mechanical parameters: Peak airway pressure (Paw peak) and plateau pressure (Paw plateau).

         • Occurrence of intraoperative pulmonary adverse effects
         * Occurrence of intraoperative desaturation (spo2 <92%) or change in heart rate and arterial blood pressure by at least 15% of baseline values

      <!-- -->

      1. Sample size Based on the primary outcome, sample size calculation was done using the comparison of incidence of lung collapse between standard ventilation and a lung recruitment manoeuver in pediatric patients scheduled for abdominal laparoscopic surgery using a four point aeration score by ultrasound imaging.

         Calculation was done based on comparing 2 proportions from independent samples in a prospective study using Chi test, the α-error level was fixed at 0.05, the power was set at 80% and the intervention groups ratio was set at 1. As previously published (30), the incidence of lung collapse among lung recruitment manoeuver group was 45% while it was 90% in standard ventilation group. Accordingly, the minimum optimum sample size should be 16 participants in each group to detect a real difference of 10% in incidence of lung collapse. Sample size calculation was done using PS Power and Sample Size Calculations software, version 3.0.11 for MS Windows (William D. Dupont and Walton D., Vanderbilt University, Nashville, Tennessee, USA).
      2. Statistical Analysis Normally distributed numerical data will be statistically described in terms of mean , standard deviation (SD), while not-normal data will be represented as median and range or inter-quartile range (IQR). Qualitative (categorical) data will be described in frequencies (number of cases) and percentage. Numerical data will be tested for the normal assumption using Kolmogorov Smirnov test.

         Comparison of numerical variables between the study groups will be done using Student t test for independent samples in comparing normally distributed data and Mann Whitney U test for independent samples when data are not normally distributed. For comparing categorical data, Chi-square test will be performed. Exact test will be used instead when the expected frequency is less than 5. A probability value (p value) less than 0.05 is considered statistically significant. All statistical calculations will be done using computer programs Microsoft Excel 2007 (Microsoft Corporation, NY, USA) and IBM SPSS (Statistical Package for the Social Science; IBM Corp, Armonk, NY, USA) release 22 for Microsoft Windows.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Parental Consent
* Scheduled for undergoing abdominal laparoscopic surgery
* American Society of Anaesthesiologists (ASA) physical status classification Ⅰ-Ⅱ

Exclusion Criteria:

* Emergency and thoracic procedures
* Significant pre-existing pulmonary, cardiac or chest wall diseases
* Abdominal distension
* Acute airway infection
* Previous thoracic procedure

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
The lung aeration score by ultrasound | from start of surgery till half an hour postoperative
  Four Lung ultrasound patterns were defined according to the degree of B lines: (0) fewer than three isolated B lines; (1) multiple well defined B lines; (2) multiple coalescent B lines and (3) white lung. The sum of the points obtained in all the 12 lung areas will constitute the lung aeration score, ranging from 0-36 for the whole thorax. This score is inversely proportional to the degree of lung aeration and directly proportional to the degree of lung atelectasis.

SECONDARY OUTCOMES:
Incidence of hemodynamic instability or oxygen desaturation | from start of surgery till half an hour postoperative
  with the sustained inflation recruitment manoeuver

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forgiarini Junior LA, Esquinas AM. [Atelectasis in postoperative bariatric surgery: how many understand them?]. Braz J Anesthesiol. 2018 Jan-Feb;68(1):109-110. doi: 10.1016/j.bjan.2017.01.004. Epub 2017 May 24. No abstract available. PMID 28551061
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Malbrain ML, De Laet I, De Waele JJ, Sugrue M, Schachtrupp A, Duchesne J, Van Ramshorst G, De Keulenaer B, Kirkpatrick AW, Ahmadi-Noorbakhsh S, Mulier J, Pelosi P, Ivatury R, Pracca F, David M, Roberts DJ. The role of abdominal compliance, the neglected parameter in critically ill patients - a consensus review of 16. Part 2: measurement techniques and management recommendations. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):406-32. doi: 10.5603/AIT.2014.0063. PMID 25432559
- [Background] Yang D, Grant MC, Stone A, Wu CL, Wick EC. A Meta-analysis of Intraoperative Ventilation Strategies to Prevent Pulmonary Complications: Is Low Tidal Volume Alone Sufficient to Protect Healthy Lungs? Ann Surg. 2016 May;263(5):881-7. doi: 10.1097/SLA.0000000000001443. PMID 26720429